CLINICAL TRIAL: NCT05101135
Title: This Study Evaluates the Addition of Dapagliflozin in the Treatment of Type 2 Diates With Metformin and JT-001 Combination Therapy.
Brief Title: To Evaluate the Efficacy and Safety of JT-001 add-on in Paatients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin and Dapagliflozin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JLP-2008-301
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — GS-621763

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JT-001 (Experimental): Drug: JT-001
  Interventions: Drug: JT-001
- JT-001 Placebo (Placebo Comparator): Drug: JT-001 Placebo
  Interventions: Drug: JT-001 Placebo

INTERVENTIONS:
Drug: JT-001 — Subjects take the investigational products once a day for 24 weeks.
  Arms: JT-001
Drug: JT-001 Placebo — Subjects take the investigational products once a day for 24 weeks.
  Arms: JT-001 Placebo

SUMMARY:
A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase III Study to Evaluate the Efficacy and Safety of JT-001 Add-on in Patients with Type 2 Diabetes Mellitus Inadequately Controlled with Metformin and Dapagliflozin.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years or older with type 2 diabetes mellitus
2. Subjects with 7.0% ≤ HbA1c ≤ 11% at baseline
3. Those with > 45 kg/m2 of BMI
4. Those who voluntarily signed the informed consent to participate in this study

Exclusion Criteria:

1. Those who had allergic reaction to main ingredients or components of the investigational products.
2. Patients with the following major systemic disease

   * Patients with type 1 diabetes mellitus, secondary diabetes, or congenital renal diabetes etc.)
   * Patients with pituitary insufficiency or adrenal dysfunction
   * Patients with uncontrolled glycosemia(FPG > 270 mg/dL)
   * Patients with uncontrolled hypertension(SBP > 180 mmHg or DBP > 110 mmHg
   * Patients with severe hypertriglyceridemia (Triglyceride > 500 mg/dL)
   * Patients with severe renal dysfunction
   * Patients with liver dysfunction
   * Patients with AIDS
   * Those with clinically significant severe infection or trauma based on an investigator's judgement
   * Patients with pulmonary infarction, severe pulmonary dysfunction, hypoxemia
   * Unstable mental illness not regulated by drugs
   * Those who suffered from gastrointestinal diseases that may affect the absorption, distribution, metabolism, and excretion of investigational products or had underwent surgery;
   * Those who had genetic disorders such as galactose intolerance, Lapp lactose deficiency, or glucose-galactose malabsorption
3. Those with a history of malignant tumor within 5 years
4. Those with history of alcohol or drug abuse within 1 years
5. Those with heart failure (NYHA class II~IV) or who had suffered from heart failure within 6 months
6. Those who underwent surgery requiring general anesthesia within 4 weeks as of Visit 1 or who are scheduled to receive such surgery within 4 weeks after the study ends
7. Those who need to take prohibited concomitant medications stated during the study period.
8. Females who are pregnant or breastfeeding or patients planning to become pregnant or of childbearing potential, but not using any recognized contraceptive method
9. Those who are judged unsuitable for the study by a principal investigator or investigators
10. Those who have been administered with the following drugs or expected to require the continued administration during the study period:

    * Those who have been administered with obesity drugs within 12 weeks
    * Those being administered with thyroid medications and whose dose has been modified within 6 weeks
    * Those administered with systemic steroid agents (Prednisolone, >30 mg/day) within 2 weeks
    * Those being administered with diuretics and whose dose has been modified within 8 weeks as (however, dose reduction is accepted.)
11. Those who are currently participating in other ongoing clinical studies or those who have taken the investigational products from other clinical studies within 12 weeks

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes in HbA1c | 24th Week
  Changes in HbA1c at the 24th week from the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heo JH, Han KA, Hong JH, Seo HA, Hong EG, Yu JM, Jung HS, Cha BS. Pioglitazone as Add-on Therapy in Patients with Type 2 Diabetes Mellitus Inadequately Controlled with Dapagliflozin and Metformin: Double-Blind, Randomized, Placebo-Controlled Trial. Diabetes Metab J. 2024 Sep;48(5):937-948. doi: 10.4093/dmj.2023.0314. Epub 2024 Feb 2. PMID 38310875